CLINICAL TRIAL: NCT01276613
Title: Tissue Pharmacokinetics of Intraoperative Gemcitabine in Resectable Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Per memo from study team
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0371; NCI-2011-00244 (Registry Identifier: NCI CTRP); RSD1429) (Other Grant/Funding Number: RSNA); WS#23 (Other Grant/Funding Number: GE)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
Keywords: Resectable Adenocarcinoma of the Pancreas; Gemcitabine; Gemcitabine Hydrochloride; Gemzar
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intraoperative Gemcitabine (Experimental): Gemcitabine administered by the anesthesiologist as a dose of 1,000mg/m2 at a fixed dose rate of 10mg/m2/min. Drug infusion started 100 minutes prior to complete gross tumor removal in order to have drug administration complete at tumor removal.
  Interventions: Drug: Gemcitabine
- Intraoperative Gemcitabine + Losartan (Experimental): Losartan 50 mg by mouth daily for one week and 50 to 100 mg of Losartan by mouth daily for at least 1 week and at most 3 weeks prior to surgical resection.
  Gemcitabine administered by the anesthesiologist as a dose of 1,000mg/m2 at a fixed dose rate of 10mg/m2/min. Drug infusion started 100 minutes prior to complete gross tumor removal in order to have drug administration complete at tumor removal.
  Interventions: Drug: Gemcitabine; Drug: Losartan

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine administered by the anesthesiologist as a dose of 1,000mg/m2 at a fixed dose rate of 10mg/m2/min.
  Other Names: Gemcitabine Hydrochloride; Gemzar
Drug: Losartan — 50 mg by mouth daily for one week and 50 to 100 mg of Losartan by mouth daily for at least 1 week and at most 3 weeks prior to surgical resection.
  Arms: Intraoperative Gemcitabine + Losartan

SUMMARY:
The goal of this clinical research study is to learn if gemcitabine can enter pancreas cancer cells, to measure the amount of it that may enter the cells, and for biomarker testing. Biomarkers may be related to participant's reaction to the study drug.

DETAILED DESCRIPTION:
The Study Drugs:

Gemcitabine is a drug used to treat pancreatic cancer. However, there are no studies that show that gemcitabine is able to enter pancreatic cancer cells.

Losartan is a drug that lowers blood pressure. It also may increase the amount of gemcitabine that reaches the cancer cells. Participant may be asked to take this drug before participant's surgery.

Before Surgery:

If participant is found to be eligible and participant agrees to take part in this study, the following tests will be done before participant's surgery:

* Participant will have a routine CT (computed tomography) scan and a research MRI (magnetic resonance imaging) of participant's abdomen to check the status of the disease.
* Blood (about 3-4 teaspoons) will be drawn for biomarker testing.

Participant may be asked to take losartan for 2-4 two to four weeks before participant's surgery (described below).

Surgery:

Participant's surgery will be performed in the same way as it would be even if participant was not taking part in this study. Participant will sign a separate consent form for surgery. The length of the surgery and the time participant is under anesthesia are not changed by taking part in the study.

To measure how much gemcitabine enters pancreas cancer cells, participants who are having their pancreatic cancer removed by surgery will receive an infusion of gemcitabine during the surgery. Some of the pancreatic cancer tissue removed then will be checked to learn if gemcitabine is found in the cancer cells.

During surgery, participant will have routine procedures to learn if the disease has spread to other areas. If the disease has spread beyond the pancreas, surgical removal is not possible.

If for any reason during the surgery, the surgeon decides that removal of the pancreas is not possible, participant will not receive gemcitabine and participation in this study will end.

If there are no signs of spread or other reasons the cancer cannot be removed, the surgeon will begin the process of removal of the disease.

Gemcitabine Infusion:

Participant will receive an infusion of gemcitabine just before the surgeon begins to remove the cancer. Gemcitabine will be given through an infusion catheter that is placed in the operating room after participant is asleep. The infusion will take over 100 minutes. The infusion catheter is not required for the study but is a standard of care procedure for all participants who are having pancreatic cancer surgery. Participant will sign a separate consent form for the infusion catheter.

Losartan Administration:

If participant is asked to take losartan, participant will take 1 tablet by mouth every day for up to 4 weeks before participant's surgery. After Week 1, the study staff will tell participant if participant's dose will stay the same or increase, based on any side effects that participant may have.

Blood and Tissue Collection:

Up to 10 blood samples (about 1 tablespoon each time) will be drawn during surgery starting before the gemcitabine infusion begins and at the end of surgery. The blood samples are used to measure the levels of gemcitabine in participant's blood at different time points. This is called pharmacokinetic (PK) testing. The blood will also be used for biomarker testing. Biomarkers are chemical "markers" in the blood/tissue that may be related to participant's reaction to the study drug.

Some of the tumor tissue and normal tissue removed during surgery will be collected to learn if gemcitabine is able to enter the tissue cells and for biomarker testing.

Length of Study:

Participant's active participation in this study will be over once participant has had surgery and completed the follow-up. The research team will continue to collect information on participant for 30 days after surgery (or until participant is no longer having side effects).

Follow-Up:

The study team will follow participant's health status for 30 days after surgery to check if participant is having any side effects from gemcitabine. This follow-up will be done daily while participant is in the hospital recovering from the surgery. Follow-up will also occur at the time of a routine clinic visit, or by phone call at least once weekly. These calls should last about 5 minutes each.

This is an investigational study. Gemcitabine is FDA approved and commercially available for the treatment of pancreatic cancer. Its use during surgery is investigational.

Losartan is FDA approved and commercially available for the treatment of high blood pressure and diabetic nephropathy. It is not approved for the treatment of pancreatic cancer.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreas is required. Patients with Islet cell tumors are not eligible.
2. Patients do not have known metastases.
3. Patients must have potentially resectable pancreatic cancer and have agreed to undergo surgical resection at M D Anderson Cancer Center. They will have undergone staging (physical examination, chest x-ray, contrast enhanced CT or MRI (if CT contraindicated) and/or angiogram to determine resectability. Potentially resectable is defined as:No extra-pancreatic disease; No evidence (on CT/MRI) of tumor extension to the celiac axis or SMA; No evidence (CT/MRI or angiogram) of occlusion of the SMV or SMPV confluence.
4. Patients with a Karnofsky performance status greater than 70 are eligible.
5. There will be no upper age restriction. Patients less than 18 years of age are excluded from the protocol because adenocarcinoma of the pancreas is rarely seen in the pediatric population.
6. Adequate renal, and bone marrow function: Leukocytes >= 3,000/uL; Absolute neutrophil count >= 1,500/uL; Platelets >= 100,000/Ul; Serum creatinine <= 2.0 mg/dL.
7. Adequate Hepatic function (endoscopic or percutaneous drainage as needed): Total bilirubin < = 3 X institutional upper limits of normal (ULN); AST (SGOT)/ALT (SGPT) <= 5 X institutional ULN.
8. Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude administration of gemcitabine. Patients with uncontrolled congestive heart failure, unstable angina and myocardial infarction within 3 months will be excluded.
9. Patient is not pregnant. Women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to practice adequate contraception and to refrain from breast-feeding, as specified in the informed consent.
10. Patients must sign a study-specific consent form.

Exclusion Criteria:

1. Patient has received preoperative chemotherapy and/or radiation.
2. Major cardiovascular or pulmonary comorbidity that precludes use of general anesthesia.
3. Identification of metastatic disease.
4. Inability to comply with study and/or follow-up procedures.
5. Patients < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Intratumoral Gemcitabine Levels in Human Pancreatic Cancer Tissue | Collection during surgery, participants followed 30 days post surgery
  Pharmacokinetic (PK) Testing of up to 10 blood samples (about 1 tablespoon each time) drawn during surgery starting before gemcitabine infusion and at end of surgery. Blood samples used to measure levels of gemcitabine in blood at the different time points.
Gemcitabine DNA Levels in Human Pancreatic Cancer Tissue | Before surgery, participants followed 30 days post surgery
  CT scans analyzed, mapping 3 to 4 areas of pancreatic tumor based on differential enhancement patterns within the tumors, where each selected region is uniform within 5-10 HU at each phase of the CT. Each region will comprise no more than 33% of the greatest size of the tumor. Model parameters for each region plugged into the predictive equations for YVmax, YTmax, R0, and AUC.

SECONDARY OUTCOMES:
Effect of Losartan on Gemcitabine DNA Incorporation Human Pancreatic Cancer Tissue | Before surgery, participants followed 30 days post surgery
  Root mean square error estimated of prediction from the pre-therapy CT scan to be 0.14 pg dFdC/ng dG. From this estimate of the error of prediction, 80% power calculated to detect an absolute increase in gemcitabine delivery of 0.36 pg dFdC/ng dG and a 90% power to detect an absolute increase in gemcitabine delivery of 0.42 pg dFdC/ng dG in a given participant.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Koay EJ, Truty MJ, Cristini V, Thomas RM, Chen R, Chatterjee D, Kang Y, Bhosale PR, Tamm EP, Crane CH, Javle M, Katz MH, Gottumukkala VN, Rozner MA, Shen H, Lee JE, Wang H, Chen Y, Plunkett W, Abbruzzese JL, Wolff RA, Varadhachary GR, Ferrari M, Fleming JB. Transport properties of pancreatic cancer describe gemcitabine delivery and response. J Clin Invest. 2014 Apr;124(4):1525-36. doi: 10.1172/JCI73455. Epub 2014 Mar 10. PMID 24614108
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org